CLINICAL TRIAL: NCT02207413
Title: Safety and Immunogenicity Study of GSK Biologicals' Quadrivalent Influenza Candidate Vaccine (GSK23211381A) Manufactured With a New Process in Adults and Children
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Candidate Vaccine (GSK2321138A) Manufactured Using a New Process in Adults and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201251
Record Dates: First submitted 2014-07-24; First posted 2014-08-04 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Quadrivalent influenza vaccine; Safety; Children; Adults; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Influsplit Tetra_IP Adult Group (Experimental): Subjects in the Influsplit Tetra_IP group aged between 18 to 49 years received 1 dose of Influsplit Tetra™ vaccine produced by investigational process (IP) at Day 0. Influsplit Tetra™ vaccine produced by IP was administered intramuscularly in the deltoid region of left or non-dominant arm.
  Interventions: Biological: Influsplit Tetra™ vaccine produced by investigational process (IP)
- Influsplit Tetra_LP Adult Group (Active Comparator): Subjects in the Influsplit Tetra_LP aged between 18 to 49 years received 1 dose of Influsplit Tetra™ vaccine produced by currently licensed process (LP) at Day 0. Influsplit Tetra™ vaccine produced by currently LP was administered intramuscularly in the deltoid region of left or non-dominant arm.
  Interventions: Biological: Influsplit Tetra™ vaccine produced by licensed process (LP)
- Influsplit Tetra_IP 3-17y Group (Experimental): Subjects in the Influsplit Tetra_IP group aged between 3 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by IP at Day 0. Influsplit Tetra™ vaccine produced by IP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
  Interventions: Biological: Influsplit Tetra™ vaccine produced by investigational process (IP)
- Influsplit Tetra_LP 3-17y Group (Active Comparator): Subjects in the Influsplit Tetra_LP group aged between 3 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by LP at Day 0. Influsplit Tetra™ vaccine produced by LP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
  Interventions: Biological: Influsplit Tetra™ vaccine produced by licensed process (LP)
- Influsplit Tetra_IP 6-35m Group (Experimental): Subjects in the Influsplit Tetra_IP group aged between 6 months to 35 months received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Influsplit Tetra™ vaccine produced by IP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
  Interventions: Biological: Influsplit Tetra™ vaccine produced by investigational process (IP)
- Influsplit Tetra_LP 6-35m Group (Active Comparator): Subjects in the Influsplit Tetra_LP group aged between 6 months to 35 months received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Influsplit Tetra™ vaccine produced by LP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
  Interventions: Biological: Influsplit Tetra™ vaccine produced by licensed process (LP)

INTERVENTIONS:
Biological: Influsplit Tetra™ vaccine produced by investigational process (IP) — Influsplit Tetra™ vaccine using a new manufacturing process administered intramuscularly (IM) in the deltoid region of non-dominant arm (Dose 1) in Adults Group and in non-dominant deltoid or left anterolateral thigh (Dose 1) and dominant deltoid or right anterolateral (Dose 2 - unprimed subjects) in 6-35m and 3-17y Groups.
  Other Names: Fluarix Tetra™; Fluarix Quadrivalent® (GSK2321138A)
  Arms: Influsplit Tetra_IP 3-17y Group; Influsplit Tetra_IP 6-35m Group; Influsplit Tetra_IP Adult Group
Biological: Influsplit Tetra™ vaccine produced by licensed process (LP) — Influsplit Tetra™ vaccine using a licensed manufacturing process administered IM in the deltoid region of non-dominant arm (Dose 1) in Adults Group and in non-dominant deltoid or left anterolateral thigh (Dose 1) and dominant deltoid or right anterolateral (Dose 2 - unprimed subjects) in 6-35m and 3-17y Groups.
  Other Names: Fluarix Tetra™; Fluarix Quadrivalent® (GSK2321138A)
  Arms: Influsplit Tetra_LP 3-17y Group; Influsplit Tetra_LP 6-35m Group; Influsplit Tetra_LP Adult Group

SUMMARY:
The purpose of this trial is to demonstrate the acceptable safety profile and the immunological non-inferiority of the FLU D-QIV vaccine manufactured with this investigational process (FLU D-QIV Investigational Process [IP]) compared to FLU D-QIV manufactured with the current licensed process (FLU D-QIV Licensed Process [LP]).

DETAILED DESCRIPTION:
This study will enroll 3 age cohorts:

Adults: 18-49 years, Children: 3-17 years and 6-35 months of age.

ELIGIBILITY:
Inclusion Criteria:

Adults 18-49 years cohort:

* A male or female between, and including, 18 and 49 years of age at the time of vaccination.
* Subjects who the investigator believes that they/their parent(s)/Legally Acceptable Representatives (LAR(s)) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/parent(s)/LAR(s) of the subject.
* Written informed assent obtained from the subject if/as required by local regulations.
* Healthy subjects or those with chronic well-controlled disease as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception for 2 months after vaccination.

Pediatric cohort:

United States:

• A male or female subject between, and including, the ages of 3 and 17 years in the United States.

Rest of the World:

• A male or female subject between, and including, the ages of 6 months to 17 years all countries with the exception of the United States.

All participating countries:

* Subjects who the investigator believes that they/their parent(s)/Legally Acceptable Representatives (LAR(s)) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/parent(s)/LAR(s) of the subject.
* Written informed assent obtained from the subject if/as required by local regulations.
* Healthy subjects or those with chronic well-controlled disease as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

Adults aged 18-49 years cohort:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical or device).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Any administration of a long-acting immune-modifying drug within 6 months before study start, or planned administration during the study period.
* Administration of an influenza vaccine during the 6 months preceding entry into the study.
* Administration of a vaccine not foreseen by the study protocol within 30 days before vaccination or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Acute or un-controlled, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Any history of Guillain-Barré Syndrome.
* Acute disease and/or fever at the time of enrolment. Fever is defined as temperature ≥ 38.0ºC/100.4ºF.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any contra-indication to intramuscular administration of influenza vaccines.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Pediatric cohort

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical or device).
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccination dose. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Any administration of a long-acting immune-modifying drug within 6 months before study start, or planned administration during the study period.
* Administration of an influenza vaccine during the 6 months preceding entry into the study.
* Administration of a vaccine not foreseen by the study protocol within 30 days before vaccination or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Acute or un-controlled, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory tests.
* Any history of Guillain-Barré Syndrome.
* Acute disease and/or fever at the time of enrolment. Fever is defined as temperature ≥ 38.0ºC/100.4ºF.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Any contra-indication to intramuscular administration of influenza vaccines.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1886 (Actual)
Dates: Start 2014-08-18; Primary Completion 2015-04-18 (Actual); Study Completion 2015-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (4):
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
- GSK Investigational Site, Dhaka, Bangladesh
- Czechia (11):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chlumec nad Cidlinou
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Lipník nad Bečvou
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- France (7):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
- Germany (17):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Schönau am Königssee, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Neumünster
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Wroclaw
- Spain (6):
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

REFERENCES:
- [Derived] Claeys C, Drame M, Garcia-Sicilia J, Zaman K, Carmona A, Tran PM, Miranda M, Martinon-Torres F, Thollot F, Horn M, Schwarz TF, Behre U, Merino JM, Sadowska-Krawczenko I, Szymanski H, Schu P, Neumeier E, Li P, Jain VK, Innis BL. Assessment of an optimized manufacturing process for inactivated quadrivalent influenza vaccine: a phase III, randomized, double-blind, safety and immunogenicity study in children and adults. BMC Infect Dis. 2018 Apr 18;18(1):186. doi: 10.1186/s12879-018-3079-8. PMID 29669531

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primed subjects: Received 2 doses of seasonal influenza vaccine separated by at least one month during the last season or had received at least 1 dose prior to last season. Unprimed subjects: Did not receive any seasonal influenza vaccine in the past or received only 1 dose for the first time in the last influenza season.
Pre-assignment Details: For 5 subjects, study vaccine dose not administered at all but subject number was allocated.
  Some data has been analysed in sub-groups by age: 3-4 years, 5-17 years, 6 months to <5 years.
Period: Overall Study
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Started | 60 | 60 | 410 | 411 | 466 | 474
Completed | 59 | 60 | 410 (Primed subjects: 309; Unprimed subjects: 101) | 410 (Primed subjects: 312; Unprimed subjects: 98) | 459 (Primed subjects: 40; Unprimed subjects: 419) | 461 (Primed subjects: 41; Unprimed subjects: 420)
Not Completed | 1 | 0 | 0 | 1 | 7 | 13
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 3 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group | Total
Number analyzed (Participants) | 60 | 60 | 410 | 411 | 466 | 474 | 1881
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.8 (8.7) | 31.2 (9.3) | 9.4 (4.2) | 9.4 (4.2) | NA (NA) — Calculated in 'months' as per group definition. | NA (NA) — Calculated in 'months' as per group definition. | 12.1 (8.67)
Age, Continuous [Mean (Standard Deviation); unit: Months] | NA (NA) — Calculated in 'years' as per group definition. | NA (NA) — Calculated in 'years' as per group definition. | NA (NA) — Calculated in 'years' as per group definition. | NA (NA) — Calculated in 'years' as per group definition. | 19.7 (8.0) | 19.9 (8.3) | 19.8 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 35 | 196 | 187 | 223 | 209 | 891
  Male | 19 | 25 | 214 | 224 | 243 | 265 | 990

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Aged 18-49 Years Reporting Solicited Local Adverse Events (AEs).
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain = significant pain at rest and pain that prevented normal everyday activities. Grade 3 redness and swelling = greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Adult-Total Vaccinated cohort which included all subjects aged 18 to 49 years with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Pain | 41 | 32
  Grade 3 Pain | 1 | 0
  Any Redness | 1 | 1
  Grade 3 Redness | 0 | 0
  Any Swelling | 2 | 4
  Grade 3 Swelling | 0 | 0

2. Primary Outcome: Number of Subjects Aged 18-49 Years Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue,gastrointestinal symptoms, headache, Joint Pain, myalgia, shivering and fever. Gastrointestinal symptoms included nausea, vomiting, diarrhoea and/or abdominal pain. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Grade 3 was defined as symptoms that prevented normal activities. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Any fever was defined as subjects with a documented temperature of greater than or equal to (≥) 38°C/100.4°F by any route and all subjects reporting temperature less than (< )38°C but with missing values (MC) for at least one day during the solicited period. Grade 3 fever was defined as temperature ≥39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Fatigue | 32 | 20
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 28 | 20
  Any Gastrointestinal symptoms | 6 | 6
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 4 | 4
  Any Headache | 30 | 16
  Grade 3 Headache | 1 | 1
  Related Headache | 26 | 14
  Any Joint Pain | 8 | 5
  Grade 3 Joint Pain | 0 | 0
  Related Joint Pain | 8 | 5
  Any Myalgia | 21 | 13
  Grade 3 Myalgia | 1 | 0
  Related Myalgia | 20 | 13
  Any Shivering | 9 | 7
  Grade 3 Shivering | 1 | 0
  Related Shivering | 8 | 6
  Any Fever | 2 | 2
  Fever (≥38.0°C) | 2 | 1
  Grade 3 Fever | 0 | 0
  Related Fever | 2 | 2
  ≥38.0°C Related Fever | 2 | 1

3. Primary Outcome: Duration of Solicited Local and General AEs in Subjects Aged 18-49 Years.
Description: Duration was defined as number of days with any grade of local and general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Adult-Total Vaccinated cohort which included all subjects aged 18 to 49 years with at least one vaccine administration documented.
  N = Number of subjects with the symptom and without the missing confirmed grade
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 41 | 32
Days
  Fatigue: number analyzed (Participants) | 32 | 20
  Fatigue | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 6 | 6
  Gastrointestinal symptoms | 1.5 [1.0 to 4.0] | 1.0 [1.0 to 3.0]
  Headache: number analyzed (Participants) | 30 | 16
  Headache | 1.0 [1.0 to 6.0] | 1.5 [1.0 to 5.0]
  Joint Pain: number analyzed (Participants) | 8 | 5
  Joint Pain | 1.0 [1.0 to 4.0] | 3.0 [1.0 to 4.0]
  Myalgia: number analyzed (Participants) | 21 | 13
  Myalgia | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0]
  Pain | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 7.0]
  Redness: number analyzed (Participants) | 1 | 1
  Redness | 2.0 [2.0 to 2.0] | 1.0 [1.0 to 1.0]
  Shivering: number analyzed (Participants) | 9 | 7
  Shivering | 2.0 [1.0 to 4.0] | 3.0 [1.0 to 5.0]
  Swelling: number analyzed (Participants) | 2 | 4
  Swelling | 1.5 [1.0 to 2.0] | 2.5 [2.0 to 4.0]
  Fever: number analyzed (Participants) | 2 | 2
  Fever | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]

4. Primary Outcome: Number of Subjects Aged 18-49 Years Reporting Solicited Oculorespiratory Syndrome (ORS) Like Symptoms.
Description: Oculorespiratory syndrome (ORS) was defined as the occurrence within 24 hours after vaccination of one or more of the following newly onset symptoms: bilateral red eyes, cough, wheeze, chest tightness, difficulty breathing, difficulty swallowing, hoarseness, sore throat, facial swelling. Any was defined as any ORS symptom regardless of intensity grade or relationship to vaccination. Grade 3 ORS was defined as ORS symptoms that prevented normal activities. Related ORS was defined as ORS symptom(s) assessed by the investigator as causally related to the vaccination.
Time Frame: During the 3-day (Days 0-2) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 59
Subjects
  Any Chest Tightness | 0 | 0
  Grade 3 Chest Tightness | 0 | 0
  Related Chest Tightness | 0 | 0
  Any Cough | 3 | 2
  Grade 3 Cough | 0 | 0
  Related Cough | 3 | 1
  Any Difficulty Breathing | 0 | 0
  Grade 3 Difficulty Breathing | 0 | 0
  Related Difficulty Breathing | 0 | 0
  Any Hoarseness | 1 | 1
  Grade 3 Hoarseness | 0 | 0
  Related Hoarseness | 1 | 1
  Any Red Eyes | 1 | 1
  Grade 3 Red Eyes | 0 | 0
  Related Red Eyes | 1 | 0
  Any Sore Throat | 4 | 2
  Grade 3 Sore Throat | 0 | 0
  Related Sore Throat | 3 | 1
  Any Swallowing Difficulty | 3 | 1
  Grade 3 Swallowing Difficulty | 0 | 0
  Related Swallowing Difficulty | 2 | 0
  Any Swelling of the face | 0 | 0
  Grade 3 Swelling of the face | 0 | 0
  Related Swelling of the face | 0 | 0
  Any Wheezing | 0 | 0
  Grade 3 Wheezing | 0 | 0
  Related Wheezing | 0 | 0

5. Primary Outcome: Number of Subjects Aged 18-49 Years Reporting the Occurrence of Medically Attended Events (MAEs).
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s). Grade 3 was defined as MAE that prevented normal activities. Related was defined as MAE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (approximately 21 days following vaccination)
Population: The analysis was performed on the Adult-Total Vaccinated cohort which included all subjects aged 18 to 49 years with at least one vaccine administration documented.
  1 subject withdrew consent in the Influsplit Tetra_LP Adult Group and did not complete the study but was administered a study vaccine dose.
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any MAE(s) | 9 | 8
  Grade 3 MAE(s) | 3 | 1
  Related MAE(s) | 0 | 0

6. Primary Outcome: Number of Subjects Aged 3-17 Years Reporting Solicited Local Adverse Events (AEs).
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain = Cried when limb was moved/spontaneously painful. Grade 3 redness and swelling = greater than 50 millimeters (mm) i.e. >50mm.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 3 to 17 years, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 410 | 410
Subjects
  Any Pain, Dose 1 | 243 | 253
  Grade 3 Pain, Dose 1 | 14 | 20
  Any Redness, Dose 1 | 118 | 119
  Grade 3 Redness, Dose 1 | 8 | 7
  Any Swelling, Dose 1 | 102 | 100
  Grade 3 Swelling, Dose 1 | 7 | 7
  Any Pain, Dose 2: number analyzed (Participants) | 103 | 99
  Any Pain, Dose 2 | 36 | 39
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Pain, Dose 2 | 0 | 2
  Any Redness, Dose 2: number analyzed (Participants) | 103 | 99
  Any Redness, Dose 2 | 25 | 21
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 103 | 99
  Any Swelling, Dose 2 | 16 | 17
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Swelling, Dose 2 | 1 | 0
  Any Pain, Across Doses | 252 | 264
  Grade 3 Pain, Across Doses | 14 | 21
  Any Redness, Across Doses | 129 | 128
  Grade 3 Redness, Across Doses | 8 | 7
  Any Swelling, Across Doses | 109 | 110
  Grade 3 Swelling, Across Doses | 8 | 7

7. Primary Outcome: Number of Subjects Aged 3-4 Years Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were drowsiness, irritability/fussiness, loss of appetite and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 irritability/fussiness was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Grade 3 drowsiness was defined as drowsiness that prevented normal activity. Any fever was defined as subjects with a documented temperature of greater than or equal to (≥) 38°C/100.4°F by any route and all subjects reporting temperature less than (< )38°C but with missing values (MC) for at least one day during the solicited period. Grade 3 fever was defined as temperature greater than (>) 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 3 to 4 years, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Groups:
- Influsplit Tetra_IP 3-4y Group: Subjects in the Influsplit Tetra_IP group aged between 3 to 4 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Influsplit Tetra™ vaccine produced by IP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
- Influsplit Tetra_LP 3-4y Group: Subjects in the Influsplit Tetra_LP group aged between 3 to 4 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Influsplit Tetra™ vaccine produced by LP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
Arm/Group | Influsplit Tetra_IP 3-4y Group | Influsplit Tetra_LP 3-4y Group
Number analyzed (Participants) | 70 | 72
Subjects
  Any Drowsiness, Dose 1 | 14 | 7
  Grade 3 Drowsiness, Dose 1 | 0 | 1
  Related Drowsiness, Dose 1 | 10 | 4
  Any Irritability, Dose 1 | 9 | 12
  Grade 3 Irritability, Dose 1 | 1 | 1
  Related Irritability, Dose 1 | 6 | 8
  Any Loss of appetite, Dose 1 | 9 | 14
  Grade 3 Loss of appetite, Dose 1 | 2 | 1
  Related Loss of appetite, Dose 1 | 6 | 6
  Any Fever, Dose 1 | 5 | 7
  Fever (≥38.0°C), Dose 1 | 4 | 7
  Grade 3 Fever, Dose 1 | 1 | 3
  Related Fever, Dose 1 | 1 | 5
  ≥38.0°C Related Fever, Dose 1 | 1 | 5
  Any Drowsiness, Dose 2: number analyzed (Participants) | 40 | 41
  Any Drowsiness, Dose 2 | 5 | 6
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 40 | 41
  Grade 3 Drowsiness, Dose 2 | 0 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 40 | 41
  Related Drowsiness, Dose 2 | 3 | 4
  Any Irritability, Dose 2: number analyzed (Participants) | 40 | 41
  Any Irritability, Dose 2 | 2 | 8
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 40 | 41
  Grade 3 Irritability, Dose 2 | 0 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 40 | 41
  Related Irritability, Dose 2 | 2 | 6
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 40 | 41
  Any Loss of appetite, Dose 2 | 4 | 6
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 40 | 41
  Grade 3 Loss of appetite, Dose 2 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 40 | 41
  Related Loss of appetite, Dose 2 | 2 | 3
  Any Fever, Dose 2: number analyzed (Participants) | 40 | 41
  Any Fever, Dose 2 | 0 | 4
  Fever (≥38.0°C), Dose 2]: number analyzed (Participants) | 40 | 41
  Fever (≥38.0°C), Dose 2] | 0 | 3
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 40 | 41
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 40 | 41
  Related Fever, Dose 2 | 0 | 2
  ≥38.0°C Related Fever, Dose 2: number analyzed (Participants) | 40 | 41
  ≥38.0°C Related Fever, Dose 2 | 0 | 1
  Any Drowsiness, Across Doses | 16 | 11
  Grade 3 Drowsiness, Across Doses | 0 | 2
  Related Drowsiness, Across Doses | 10 | 8
  Any Irritability, Across Doses | 10 | 16
  Grade 3 Irritability ,Across Doses | 1 | 1
  Related Irritability, Across Doses | 7 | 11
  Any Loss of appetite,Across Doses | 13 | 16
  Grade 3 Loss of appetite, Across Doses | 2 | 1
  Related Loss of appetite, Across Doses | 8 | 8
  Any Fever, Across Doses | 5 | 10
  Fever (≥38.0°C), Across Doses | 4 | 9
  Grade 3 Fever, Across Doses | 1 | 3
  Related Fever, Across Doses | 1 | 6
  ≥38.0°C Related Fever, Across Doses | 1 | 5

8. Primary Outcome: Number of Subjects Aged 5-17 Years Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache, joint pain, myalgia, shivering and fever (Fever = temperature above 38.0 degrees Celsius (°C)). Gastrointestinal symptoms included nausea, vomiting, diarrhoea and/or abdominal pain. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Any fever = all subjects with a documented temperature of ≥ 38°C/100.4°F by any route and all subjects reporting temperature < 38°C but with missing values (MC) for at least one day during the solicited period. Grade 3 fever = temperature above 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 5 to 17 years, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Groups:
- Influsplit Tetra_IP 5-17y Group: Subjects in the Influsplit Tetra_IP group aged between 5 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by IP at Day 0. Influsplit Tetra™ vaccine produced by IP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
- Influsplit Tetra_LP 5-17y Group: Subjects in the Influsplit Tetra_LP group aged between 5 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by LP at Day 0. Influsplit Tetra™ vaccine produced by LP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
Arm/Group | Influsplit Tetra_IP 5-17y Group | Influsplit Tetra_LP 5-17y Group
Number analyzed (Participants) | 340 | 338
Subjects
  Any Fatigue, Dose 1 | 94 | 99
  Grade 3 Fatigue, Dose 1 | 8 | 13
  Related Fatigue, Dose 1 | 65 | 70
  Any Gastrointestinal, Dose 1 | 35 | 32
  Grade 3 Gastrointestinal, Dose 1 | 2 | 1
  Related Gastrointestinal, Dose 1 | 18 | 16
  Any Headache, Dose 1 | 82 | 76
  Grade 3 Headache, Dose 1 | 3 | 9
  Related Headache, Dose 1 | 46 | 50
  Any Joint Pain, Dose 1 | 34 | 38
  Grade 3 Joint Pain, Dose 1 | 3 | 2
  Related Joint Pain, Dose 1 | 25 | 29
  Any Myalgia, Dose 1 | 70 | 84
  Grade 3 Myalgia, Dose 1 | 3 | 5
  Related Myalgia, Dose 1 | 55 | 72
  Any Shivering, Dose 1 | 20 | 29
  Grade 3 Shivering, Dose 1 | 0 | 3
  Related Shivering, Dose 1 | 16 | 20
  Any Fever, Dose 1 | 12 | 9
  Fever (≥38.0°C), Dose 1 | 11 | 8
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 10 | 7
  ≥38.0°C Related Fever, Dose 1 | 9 | 6
  Any Fatigue, Dose 2: number analyzed (Participants) | 63 | 58
  Any Fatigue, Dose 2 | 8 | 4
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Fatigue, Dose 2 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 63 | 58
  Related Fatigue, Dose 2 | 4 | 4
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 63 | 58
  Any Gastrointestinal, Dose 2 | 3 | 1
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 63 | 58
  Related Gastrointestinal, Dose 2 | 0 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 63 | 58
  Any Headache, Dose 2 | 2 | 7
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Headache, Dose 2 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 63 | 58
  Related Headache, Dose 2 | 2 | 4
  Any Joint Pain, Dose 2: number analyzed (Participants) | 63 | 58
  Any Joint Pain, Dose 2 | 2 | 4
  Grade 3 Joint Pain, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Joint Pain, Dose 2 | 1 | 0
  Related Joint Pain, Dose 2: number analyzed (Participants) | 63 | 58
  Related Joint Pain, Dose 2 | 1 | 3
  Any Myalgia, Dose 2: number analyzed (Participants) | 63 | 58
  Any Myalgia, Dose 2 | 3 | 9
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Myalgia, Dose 2 | 1 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 63 | 58
  Related Myalgia, Dose 2 | 2 | 7
  Any Shivering, Dose 2: number analyzed (Participants) | 63 | 58
  Any Shivering, Dose 2 | 2 | 2
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 63 | 58
  Related Shivering, Dose 2 | 0 | 1
  Any Fever, Dose 2: number analyzed (Participants) | 63 | 58
  Any Fever, Dose 2 | 3 | 0
  Fever (≥38.0°C), Dose 2: number analyzed (Participants) | 63 | 58
  Fever (≥38.0°C), Dose 2 | 2 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 63 | 58
  Grade 3 Fever, Dose 2 | 1 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 63 | 58
  Related Fever, Dose 2 | 2 | 0
  ≥38.0°C Related Fever, Dose 2: number analyzed (Participants) | 63 | 58
  ≥38.0°C Related Fever, Dose 2 | 1 | 0
  Any Fatigue, Across Doses | 97 | 101
  Grade 3 Fatigue, Across Doses | 8 | 13
  Related Fatigue, Across Doses | 66 | 72
  Any Gastrointestinal, Across Doses | 38 | 32
  Grade 3 Gastrointestinal, Across Doses | 2 | 1
  Related Gastrointestinal, Across Doses | 18 | 16
  Any Headache, Across Doses | 83 | 80
  Grade 3 Headache, Across Doses | 3 | 9
  Related Headache, Across Doses | 48 | 53
  Any Joint Pain, Across Doses | 35 | 42
  Grade 3 Joint Pain, Across Doses | 4 | 2
  Related Joint Pain, Across Doses | 25 | 32
  Any Myalgia, Across Doses | 71 | 88
  Grade 3 Myalgia, Across Doses | 4 | 5
  Related Myalgia, Across Doses | 56 | 76
  Any Shivering, Across Doses | 21 | 31
  Grade 3 Shivering, Across Doses | 0 | 3
  Related Shivering, Across Doses | 16 | 21
  Any Fever, Across Doses | 14 | 9
  Fever (≥38.0°C), Across Doses | 12 | 8
  Grade 3 Fever, Across Doses | 1 | 0
  Related Fever, Across Doses | 12 | 7
  ≥38.0°C Related Fever, Across Doses | 10 | 6

9. Primary Outcome: Duration of Solicited Local AEs in Subjects Aged 3-17 Years.
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 243 | 253
Days
  Pain, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Pain, Dose 2: number analyzed (Participants) | 36 | 39
  Pain, Dose 2 | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 3.0]
  Redness, Dose 1: number analyzed (Participants) | 118 | 119
  Redness, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Redness, Dose 2: number analyzed (Participants) | 25 | 21
  Redness, Dose 2 | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0]
  Swelling, Dose 1: number analyzed (Participants) | 102 | 100
  Swelling, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Swelling, Dose 2: number analyzed (Participants) | 16 | 17
  Swelling, Dose 2 | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 7.0]

10. Primary Outcome: Duration of Solicited General AEs in Subjects Aged 3-4 Years.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP 3-4y Group | Influsplit Tetra_LP 3-4y Group
Number analyzed (Participants) | 14 | 14
Days
  Drowsiness, Dose 1: number analyzed (Participants) | 14 | 7
  Drowsiness, Dose 1 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 7.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 5 | 6
  Drowsiness, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 5.0]
  Irritability, Dose 1: number analyzed (Participants) | 9 | 12
  Irritability, Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 4.0]
  Irritability, Dose 2: number analyzed (Participants) | 2 | 8
  Irritability, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 7.0]
  Loss of appetite, Dose 1: number analyzed (Participants) | 9 | 14
  Loss of appetite, Dose 1 | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of appetite, Dose 2: number analyzed (Participants) | 4 | 6
  Loss of appetite, Dose 2 | 1.0 [1.0 to 2.0] | 4.0 [1.0 to 7.0]
  Fever, Dose 1: number analyzed (Participants) | 5 | 7
  Fever, Dose 1 | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0]
  Fever, Dose 2: number analyzed (Participants) | 14 | 4
  Fever, Dose 2 | NA [NA to NA] — No subjects with symptom and without the missing confirmed grade were reported in this group. | 1.5 [1.0 to 3.0]

11. Primary Outcome: Duration of Solicited General AEs in Subjects Aged 5-17 Years.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 8
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP 5-17y Group | Influsplit Tetra_LP 5-17y Group
Number analyzed (Participants) | 94 | 99
Days
  Fatigue, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Fatigue, Dose 2: number analyzed (Participants) | 8 | 4
  Fatigue, Dose 2 | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0]
  Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 35 | 32
  Gastrointestinal symptoms, Dose 1 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 3 | 1
  Gastrointestinal symptoms, Dose 2 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Headache, Dose 1: number analyzed (Participants) | 82 | 76
  Headache, Dose 1 | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Headache, Dose 2: number analyzed (Participants) | 2 | 7
  Headache, Dose 2 | 2.5 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint Pain, Dose 1: number analyzed (Participants) | 34 | 38
  Joint Pain, Dose 1 | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 5.0]
  Joint Pain, Dose 2: number analyzed (Participants) | 2 | 4
  Joint Pain, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Myalgia, Dose 1: number analyzed (Participants) | 70 | 84
  Myalgia, Dose 1 | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0]
  Myalgia, Dose 2: number analyzed (Participants) | 3 | 9
  Myalgia, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Shivering, Dose 1: number analyzed (Participants) | 20 | 29
  Shivering, Dose 1 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0]
  Shivering, Dose 2: number analyzed (Participants) | 2 | 2
  Shivering, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Fever, Dose 1: number analyzed (Participants) | 12 | 9
  Fever, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 6.0]
  Fever, Dose 2: number analyzed (Participants) | 3 | 99
  Fever, Dose 2 | 2.0 [1.0 to 2.0] | NA [NA to NA] — No subjects with symptom and without the missing confirmed grade were reported in this group.

12. Primary Outcome: Number of Subjects Aged 3-17 Years Reporting Solicited Oculorespiratory Syndrome (ORS) Like Symptoms.
Description: Oculorespiratory syndrome (ORS) was defined as the occurrence within 24 hours after vaccination of one or more of the following newly onset symptoms: bilateral red eyes, cough, wheeze, chest tightness, difficulty breathing, difficulty swallowing, hoarseness, sore throat, facial swelling.
  Any = occurrence of any ORS symptom regardless of intensity grade or relationship to vaccination. Grade 3 = ORS symptoms that prevented normal activities. Related = ORS symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 3-day (Days 0-2) post-vaccination period
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 410 | 410
Subjects
  Any Chest Tightness, Dose 1 | 2 | 6
  Grade 3 Chest Tightness, Dose 1 | 0 | 0
  Related Chest Tightness, Dose 1 | 0 | 3
  Any Cough, Dose 1 | 35 | 31
  Grade 3 Cough, Dose 1 | 2 | 1
  Related Cough, Dose 1 | 12 | 10
  Any Difficulty Breathing, Dose 1 | 5 | 11
  Grade 3 Difficulty Breathing, Dose 1 | 0 | 0
  Related Difficulty Breathing, Dose 1 | 2 | 7
  Any Hoarseness, Dose 1 | 10 | 12
  Grade 3 Hoarseness, Dose 1 | 0 | 0
  Related Hoarseness, Dose 1 | 2 | 6
  Any Red Eyes, Dose 1 | 14 | 12
  Grade 3 Red Eyes, Dose 1 | 0 | 0
  Related Red Eyes, Dose 1 | 6 | 9
  Any Sore throat, Dose 1 | 14 | 18
  Grade 3 Sore throat, Dose 1 | 1 | 0
  Related Sore throat, Dose 1 | 2 | 9
  Any Swallowing Difficulty, Dose 1 | 5 | 6
  Grade 3 Swallowing Difficulty, Dose 1 | 0 | 0
  Related Swallowing Difficulty, Dose 1 | 1 | 3
  Any Swelling of the face, Dose 1 | 3 | 2
  Grade 3 Swelling of the face, Dose 1 | 0 | 0
  Related Swelling of the face, Dose 1 | 3 | 2
  Any Wheezing, Dose 1 | 1 | 5
  Grade 3 Wheezing, Dose 1 | 0 | 0
  Related Wheezing, Dose 1 | 1 | 4
  Any Chest Tightness, Dose 2: number analyzed (Participants) | 103 | 99
  Any Chest Tightness, Dose 2 | 0 | 0
  Grade 3 Chest Tightness, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Chest Tightness, Dose 2 | 0 | 0
  Related Chest Tightness, Dose 2: number analyzed (Participants) | 103 | 99
  Related Chest Tightness, Dose 2 | 0 | 0
  Any Cough, Dose 2: number analyzed (Participants) | 103 | 99
  Any Cough, Dose 2 | 6 | 13
  Grade 3 Cough, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Cough, Dose 2 | 0 | 2
  Related Cough, Dose 2: number analyzed (Participants) | 103 | 99
  Related Cough, Dose 2 | 1 | 1
  Any Difficulty Breathing, Dose 2: number analyzed (Participants) | 103 | 99
  Any Difficulty Breathing, Dose 2 | 0 | 2
  Grade 3 Difficulty Breathing, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Difficulty Breathing, Dose 2 | 0 | 0
  Related Difficulty Breathing, Dose 2: number analyzed (Participants) | 103 | 99
  Related Difficulty Breathing, Dose 2 | 0 | 0
  Any Hoarseness, Dose 2: number analyzed (Participants) | 103 | 99
  Any Hoarseness, Dose 2 | 2 | 3
  Grade 3 Hoarseness, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Hoarseness, Dose 2 | 0 | 0
  Related Hoarseness, Dose 2: number analyzed (Participants) | 103 | 99
  Related Hoarseness, Dose 2 | 1 | 0
  Any Red Eyes, Dose 2: number analyzed (Participants) | 103 | 99
  Any Red Eyes, Dose 2 | 0 | 1
  Grade 3 Red Eyes, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Red Eyes, Dose 2 | 0 | 1
  Related Red Eyes, Dose 2: number analyzed (Participants) | 103 | 99
  Related Red Eyes, Dose 2 | 0 | 1
  Any Sore Throat, Dose 2: number analyzed (Participants) | 103 | 99
  Any Sore Throat, Dose 2 | 2 | 3
  Grade 3 Sore Throat, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Sore Throat, Dose 2 | 0 | 1
  Related Sore Throat, Dose 2: number analyzed (Participants) | 103 | 99
  Related Sore Throat, Dose 2 | 0 | 0
  Any Swallowing Difficulty, Dose 2: number analyzed (Participants) | 103 | 99
  Any Swallowing Difficulty, Dose 2 | 2 | 1
  Grade 3 Swallowing Difficulty, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Swallowing Difficulty, Dose 2 | 0 | 1
  Related Swallowing Difficulty, Dose 2: number analyzed (Participants) | 103 | 99
  Related Swallowing Difficulty, Dose 2 | 1 | 0
  Any Swelling of the face, Dose 2: number analyzed (Participants) | 103 | 99
  Any Swelling of the face, Dose 2 | 0 | 1
  Grade 3 Swelling of the face, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Swelling of the face, Dose 2 | 0 | 0
  Related Swelling of the face, Dose 2: number analyzed (Participants) | 103 | 99
  Related Swelling of the face, Dose 2 | 0 | 0
  Any Wheezing, Dose 2: number analyzed (Participants) | 103 | 99
  Any Wheezing, Dose 2 | 0 | 2
  Grade 3 Wheezing, Dose 2: number analyzed (Participants) | 103 | 99
  Grade 3 Wheezing, Dose 2 | 0 | 0
  Related Wheezing, Dose 2: number analyzed (Participants) | 103 | 99
  Related Wheezing, Dose 2 | 0 | 0
  Any Chest Tightness, Across Doses | 2 | 6
  Grade 3 Chest Tightness, Across Doses | 0 | 0
  Related Chest Tightness, Across Doses | 0 | 3
  Any Cough, Across Doses | 39 | 39
  Grade 3 Cough, Across Doses | 2 | 3
  Related Cough, Across Doses | 13 | 11
  Any Difficulty Breathing, Across Doses | 5 | 13
  Grade 3 Difficulty Breathing, Across Doses | 0 | 0
  Related Difficulty Breathing, Across Doses | 2 | 7
  Any Hoarseness, Across Doses | 11 | 15
  Grade 3 Hoarseness, Across Doses | 0 | 0
  Related Hoarseness, Across Doses | 3 | 6
  Any Red Eyes, Across Doses | 14 | 13
  Grade 3 Red Eyes, Across Doses | 0 | 1
  Related Red Eyes, Across Doses | 6 | 10
  Any Sore Throat, Across Doses | 15 | 21
  Grade 3 Sore Throat, Across Doses | 1 | 1
  Related Sore Throat, Across Doses | 2 | 9
  Any Swallowing Difficulty, Across Doses | 6 | 7
  Grade 3 Swallowing Difficulty, Across Doses | 0 | 1
  Related Swallowing Difficulty, Across Doses | 2 | 3
  Any Swelling of the face, Across Doses | 3 | 3
  Grade 3 Swelling of the face, Across Doses | 0 | 0
  Related Swelling of the face, Across Doses | 3 | 2
  Any Wheezing, Across Doses | 1 | 7
  Grade 3 Wheezing, Across Doses | 0 | 0
  Related Wheezing, Across Doses | 1 | 4

13. Primary Outcome: Number of Subjects Aged 3-17 Years Reporting the Occurrence of All Medically Attended Events (MAEs) .
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s). Grade 3 was a MAE that prevented normal activities. Related was defined as a MAE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (approximately 28 days (primed subjects) and 56 days (unprimed subjects) following vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 410 | 411
Subjects
  Any MAE(s) | 59 | 52
  Grade 3 MAE(s) | 7 | 6
  Related MAE(s) | 2 | 0

14. Primary Outcome: Number of Subjects Aged 18-49 Years Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up period after vaccination
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Unsolicited AEs | 14 | 14
  Grade 3 Unsolicited AEs | 3 | 2
  Related Unsolicited AEs | 2 | 1

15. Primary Outcome: Number of Subjects Aged 3-17 Years Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: as for outcome 14
Time Frame: During the 28-day (Days 0-27) follow-up period after vaccination
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 6 months to 17 years, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 410 | 411
Subjects
  Any Unsolicited AEs | 83 | 86
  Grade 3 Unsolicited AEs | 12 | 8
  Related Unsolicited AEs | 10 | 7

16. Primary Outcome: Number of Subjects Aged 6-35 Months Reporting Fever ≥38ºC Across Doses.
Description: Any fever = all subjects with a documented temperature of ≥ 38°C/100.4°F by any route and all subjects reporting temperature < 38°C but with missing values (MC) for at least one day during the solicited period.
Time Frame: During 7 days (Days 0-6) post-vaccination
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 6 to 35 months, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 462 | 470
Subjects
  Any Fever | 76 | 70
  Fever (≥38°C) | 72 | 69

17. Primary Outcome: Number of Subjects Aged 18-49 Years, Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (approximately 21 days)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any SAEs | 1 | 1
  Related SAEs | 0 | 0

18. Primary Outcome: Number of Subjects Aged 3-17 Years, Reporting Any and Related Serious Adverse Events (SAEs)
Description: as for outcome 17
Time Frame: During the entire study period [approximately 28 days (primed subjects) and 56 days (unprimed subjects)]
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 410 | 411
Subjects
  Any SAEs | 1 | 0
  Related SAEs | 0 | 0

19. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects Aged 3-17 Years by Calculating Serum Antihaemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains.
Description: HI antibody titres were expressed as geometric mean titers (GMTs) and adjusted GMT ratios. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), FluA/Texas/50/2012 (H3N2), Flu B/Massachusetts/02/2012 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 28 post last vaccination
Population: Analysis was performed on the Pediatric According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects aged 3 to 17 years, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 403 | 402
Titers
  H1N1 | 698.0 [629.6 to 773.9] | 694.1 [625.8 to 769.7]
  H3N2 | 158.2 [143.7 to 174.2] | 171.4 [156.3 to 188.0]
  Yamagata | 479.0 [434.1 to 528.5] | 527.6 [475.5 to 585.3]
  Victoria | 237.6 [210.4 to 268.3] | 253.7 [222.7 to 289.1]
Statistical Analysis 1: Comparison: Influsplit Tetra_IP 3-17y Group vs Influsplit Tetra_LP 3-17y Group; The adjusted GMT of HI antibodies for H1N1 strain at post-vaccination of each vaccine, the GMT ratio of Influsplit Tetra_LP/ Influsplit Tetra_IP and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination antibody titer as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion (for each of the 4 strains): UL of the 95% CI for the GMT ratio (D-QIV_LP/ D-QIV_IP) is ≤ 1.5; ANCOVA; Adjusted GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — The GMTs were used to calculate the Adjusted GMTs, which in turn were used to calculate the Adjusted GMT ratio with 95% confidence interval (Ancova model: adjustment for baseline titer - pooled variance)
Statistical Analysis 2: Comparison: Influsplit Tetra_IP 3-17y Group vs Influsplit Tetra_LP 3-17y Group; The adjusted GMT of HI antibodies for H3N2 strain at post-vaccination of each vaccine, the GMT ratio of Influsplit Tetra_LP/Influsplit Tetra_IP and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination antibody titer as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion (for each of the 4 strains): UL of the 95% CI for the GMT ratio (Influsplit Tetra_LP/ Influsplit Tetra_IP) is ≤ 1.5; ANCOVA; Adjusted GMT Ratio = 1.05, 95% CI 2-sided [0.94 to 1.18] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Influsplit Tetra_IP 3-17y Group vs Influsplit Tetra_LP 3-17y Group; The adjusted GMT of HI antibodies for Yamagata strain at post-vaccination of each vaccine, the GMT ratio of Influsplit Tetra_LP/Influsplit Tetra_IP and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination antibody titer as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 2]; ANCOVA; Adjusted GMT Ratio = 1.03, 95% CI 2-sided [0.91 to 1.16] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 4: Comparison: Influsplit Tetra_IP 3-17y Group vs Influsplit Tetra_LP 3-17y Group; The adjusted GMT of HI antibodies for Victoria strain at post-vaccination of each vaccine, the GMT ratio of Influsplit Tetra_LP/Influsplit Tetra_IP and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination antibody titer as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 19, analysis 2]; ANCOVA; Adjusted GMT Ratio = 1.04, 95% CI 2-sided [0.90 to 1.21] — [estimate comment as in outcome 19, analysis 1]

20. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects Aged 6-35 Months by Calculating Serum Antihaemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains.
Description: as for outcome 19
Time Frame: At Day 28 post last vaccination
Population: Analysis was performed on the Pediatric According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects aged 6 to 35 months, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 432 | 427
Titers
  H1N1 | 97.5 [82.1 to 115.7] | 105.5 [88.2 to 126.1]
  H3N2 | 45.2 [39.0 to 52.3] | 59.9 [51.7 to 69.4]
  Yamagata | 100.8 [87.8 to 115.8] | 105.4 [91.8 to 121.0]
  Victoria | 32.1 [28.1 to 36.7] | 38.0 [33.2 to 43.5]
Statistical Analysis 1: Comparison: Influsplit Tetra_IP 6-35m Group vs Influsplit Tetra_LP 6-35m Group; The adjusted GMT of HI antibodies for H1N1 strain at post-vaccination of each vaccine, the GMT ratio of Influsplit Tetra_LP/Influsplit Tetra_IP and the 2-sided 95% CI on each GMT ratio were computed after fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination antibody titer as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion (for each of the 4 strains): UL of the 95% CI for the GMT ratio (Influsplit Tetra_LP/Influsplit Tetra_IP) is ≤ 1.5; ANCOVA; Adjusted GMT ratio = 1.07, 95% CI 2-sided [0.90 to 1.28]
Statistical Analysis 2: Comparison: Influsplit Tetra_IP 6-35m Group vs Influsplit Tetra_LP 6-35m Group; [analysis description as in outcome 19, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANCOVA; Adjusted GMT Ratio = 1.18, 95% CI 2-sided [1.00 to 1.39] — [estimate comment as in outcome 19, analysis 1]
Statistical Analysis 3: Comparison: Influsplit Tetra_IP 6-35m Group vs Influsplit Tetra_LP 6-35m Group; [analysis description as in outcome 19, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANCOVA; Adjusted GMT Ratio = 1.07, 95% CI 2-sided [0.91 to 1.27]
Statistical Analysis 4: Comparison: Influsplit Tetra_IP 6-35m Group vs Influsplit Tetra_LP 6-35m Group; [analysis description as in outcome 19, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 20, analysis 1]; ANCOVA; Adjusted GMT Ratio = 1.17, 95% CI 2-sided [0.99 to 1.38] — [estimate comment as in outcome 19, analysis 1]

21. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects Aged 18-49 Years by Calculating Serum Anti-haemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains
Description: HI antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/02/2012 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 0 and Day 21
Population: The analysis was performed on the Adult According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects aged 18 to 49 years, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 57 | 58
Titers
  [H1N1, Day 0] | 48.3 [33.4 to 69.7] | 53.6 [36.8 to 78.0]
  [H1N1, Day 21] | 655.7 [493.1 to 871.9] | 632.2 [498.8 to 801.3]
  [H3N2, Day 0] | 16.7 [12.6 to 22.2] | 16.0 [11.9 to 21.5]
  [H3N2, Day 21 | 80.5 [63.2 to 102.7] | 73.0 [59.0 to 90.5]
  [Yamagata, Day 0] | 133.3 [98.4 to 180.6] | 101.6 [76.2 to 135.4]
  [Yamagata, Day 21] | 591.4 [475.1 to 736.3] | 598.6 [480.9 to 745.0]
  [Victoria, Day 0] | 38.6 [29.5 to 50.5] | 34.8 [25.2 to 48.1]
  [Victoria, Day 21] | 263.4 [209.0 to 331.9] | 302.9 [244.0 to 376.1]

22. Secondary Outcome: Number of Seroconverted Subjects Aged 18-49 Years for Anti- Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
  The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/02/2012 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 57 | 57
Subjects
  H1N1 | 42 | 42
  H3N2 | 30 | 29
  Yamagata | 27 | 36
  Victoria | 36 | 40

23. Secondary Outcome: Number of Subjects Aged 18-49 Years, Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults.
  The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/02/2012 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 0 and Day 21
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 57 | 58
Subjects
  [H1N1, Day 0] | 35 | 35
  [H1N1, Day 21] | 56 | 57
  [H3N2, Day 0] | 15 | 14
  [H3N2, Day 21] | 49 | 49
  [Yamagata, Day 0] | 52 | 50
  [Yamagata, Day 21] | 57 | 57
  [Victoria, Day 0] | 34 | 32
  [Victoria, Day 21] | 57 | 57

24. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Four Vaccine Influenza Strains in Subjects Aged 18-49 Years.
Description: MGI was defined as the fold increase in serum haemagglutination inhibition (HI) GMTs post-vaccination compared to pre-vaccination (Day 0).
  The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/02/2012 (Yamagata) and Flu B/Brisbane/60/2008 (Victoria).
Time Frame: At Day 21
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group
Number analyzed (Participants) | 57 | 57
Fold increase
  H1N1 | 13.6 [8.9 to 20.8] | 11.5 [7.7 to 17.0]
  H3N2 | 4.8 [3.6 to 6.5] | 4.6 [3.6 to 5.7]
  Yamagata | 4.4 [3.3 to 6.0] | 6.0 [4.3 to 8.2]
  Victoria | 6.8 [5.0 to 9.2] | 8.6 [6.0 to 12.3]

25. Secondary Outcome: Number of Subjects Aged 5-17 Years Reporting Myalgia Across Doses.
Description: Any = occurrence of any myalgia symptom regardless of intensity grade or relationship to vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 5-17y Group | Influsplit Tetra_LP 5-17y Group
Number analyzed (Participants) | 340 | 338
Subjects | 71 | 88

26. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects Aged 3-17 Years by Calculating Serum Anti-haemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains
Description: as for outcome 21
Time Frame: At Day 0 and Day 28 post last vaccination
Population: The analysis was performed on the Pediatric According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects aged 3 to 17 years, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were avail
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 403 | 402
Titers
  [H1N1, Day 0] | 80.2 [69.2 to 93.0] | 87.7 [76.1 to 101.0]
  [H1N1, Day 28] | 698.0 [629.6 to 773.9] | 694.1 [625.8 to 769.7]
  [H3N2, Day 0] | 38.9 [34.6 to 43.8] | 41.9 [37.1 to 47.3]
  [H3N2, Day 28] | 158.2 [143.7 to 174.2] | 171.4 [156.3 to 188.0]
  [Yamagata, Day 0] | 58.1 [49.7 to 68.0] | 70.8 [60.4 to 83.0]
  [Yamagata, Day 28] | 479.0 [434.1 to 528.5] | 527.6 [475.5 to 585.3]
  [Victoria, Day 0] | 27.3 [23.8 to 31.3] | 28.8 [25.0 to 33.1]
  [Victoria, Day 28] | 237.6 [210.4 to 268.3] | 253.7 [222.7 to 289.1]

27. Secondary Outcome: Number of Seroconverted Subjects Aged 3-17 Years for Anti- Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: as for outcome 22
Time Frame: At Day 28 post last vaccination
Population: as for outcome 19
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 403 | 402
Subjects
  H1N1 | 274 | 269
  H3N2 | 192 | 183
  Yamagata | 273 | 268
  Victoria | 285 | 287

28. Secondary Outcome: Number of Subjects Aged 3-17 Years, Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: as for outcome 23
Time Frame: At Day 0 and Day 28 post last vaccination
Population: Analysis was performed on the Pediatric According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects aged 6 months to 17 years, who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 403 | 402
Subjects
  [H1N1, Day 0] | 308 | 314
  [H1N1, Day 28] | 393 | 395
  [H3N2, Day 0] | 245 | 252
  [H3N2, Day 28] | 377 | 378
  [Yamagata, Day 0] | 266 | 281
  [Yamagata, Day 28] | 396 | 395
  [Victoria, Day 0] | 192 | 195
  [Victoria, Day 28] | 375 | 374

29. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Four Vaccine Influenza Strains in Subjects Aged 3-17 Years.
Description: as for outcome 24
Time Frame: At Day 28 post last vaccination
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influsplit Tetra_IP 3-17y Group | Influsplit Tetra_LP 3-17y Group
Number analyzed (Participants) | 403 | 402
Fold increase
  H1N1 | 8.7 [7.6 to 10.0] | 7.9 [6.9 to 9.1]
  H3N2 | 4.1 [3.7 to 4.5] | 4.1 [3.7 to 4.6]
  Yamagata | 8.2 [7.2 to 9.4] | 7.4 [6.5 to 8.5]
  Victoria | 8.7 [7.7 to 9.8] | 8.8 [7.7 to 10.0]

30. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects Aged 6-35 Months by Calculating Serum Anti-haemagglutination (HA) Antibody Titers Against the 4 Vaccine Strains
Description: as for outcome 21
Time Frame: At Day 0 and Day 28 post last vaccination
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 432 | 427
Titers
  H1N1, Day 0: number analyzed (Participants) | 431 | 424
  H1N1, Day 0 | 11.1 [9.6 to 12.8] | 11.2 [9.7 to 12.9]
  H1N1, Day 28 | 97.5 [82.1 to 115.7] | 105.5 [88.2 to 126.1]
  H3N2, Day 0: number analyzed (Participants) | 431 | 423
  H3N2, Day 0 | 7.5 [6.8 to 8.2] | 8.4 [7.5 to 9.3]
  H3N2, Day 28 | 45.2 [39.0 to 52.3] | 59.9 [51.7 to 69.4]
  Yamagata, Day 0: number analyzed (Participants) | 431 | 423
  Yamagata, Day 0 | 8.3 [7.5 to 9.1] | 7.9 [7.2 to 8.6]
  Yamagata, Day 28 | 100.8 [87.8 to 115.8] | 105.4 [91.8 to 121.0]
  Victoria, Day 0: number analyzed (Participants) | 431 | 423
  Victoria, Day 0 | 5.7 [5.4 to 6.1] | 5.7 [5.4 to 6.1]
  Victoria, Day 28 | 32.1 [28.1 to 36.7] | 38.0 [33.2 to 43.5]

31. Secondary Outcome: Number of Seroconverted Subjects Aged 6-35 Months for Anti- Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: as for outcome 22
Time Frame: At Day 28 post last vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 432 | 427
Subjects
  H1N1 | 287 | 275
  H3N2 | 217 | 236
  Yamagata | 318 | 321
  Victoria | 213 | 211

32. Secondary Outcome: Number of Subjects Aged 6-35 Months, Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: as for outcome 23
Time Frame: At Day 0 and Day 28 post last vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 432 | 427
Subjects
  H1N1, Day 0: number analyzed (Participants) | 431 | 424
  H1N1, Day 0 | 84 | 83
  H1N1, Day 28 | 303 | 289
  H3N2, Day 0: number analyzed (Participants) | 431 | 423
  H3N2, Day 0 | 55 | 67
  H3N2, Day 28 | 232 | 259
  Yamagata, Day 0: number analyzed (Participants) | 431 | 423
  Yamagata, Day 0 | 53 | 49
  Yamagata, Day 28 | 329 | 331
  Victoria, Day 0: number analyzed (Participants) | 431 | 423
  Victoria, Day 0 | 17 | 16
  Victoria, Day 28 | 214 | 217

33. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Four Vaccine Influenza Strains in Subjects Aged 6-35 Months.
Description: as for outcome 24
Time Frame: At Day 28 post last vaccination
Population: as for outcome 28
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 432 | 427
Fold increase
  H1N1 | 8.8 [7.8 to 10.0] | 9.5 [8.3 to 10.8]
  H3N2 | 6.0 [5.4 to 6.8] | 7.1 [6.3 to 7.9]
  Yamagata | 12.2 [10.8 to 13.8] | 13.3 [11.8 to 15.0]
  Victoria | 5.6 [5.0 to 6.3] | 6.6 [5.8 to 7.4]

34. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting Fever ≥38ºC After Dose 1 and After Dose 2.
Description: Any fever = all subjects with a documented temperature of ≥ 38°C/100.4°F by any route and all subjects reporting temperature < 38°C but with missing values (MC) for at least one day during the solicited period.
  Fever = temperature of ≥ 38°C/100.4°F by any route
Time Frame: During 7 days (Days 0-6) post-vaccination
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 462 | 470
Subjects
  Any Fever, Dose 1 | 42 | 44
  Fever (≥38°C), Dose 1 | 39 | 42
  Any Fever, Dose 2: number analyzed (Participants) | 420 | 421
  Any Fever, Dose 2 | 41 | 40
  Fever (≥38°C), Dose 2: number analyzed (Participants) | 420 | 421
  Fever (≥38°C), Dose 2 | 40 | 40

35. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting Solicited Local Adverse Events (AEs).
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain = significant pain at rest and pain that prevented normal everyday activities. Grade 3 redness and swelling = greater than 50 millimeters (mm) i.e. > 50mm.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 462 | 470
Subjects
  Any Pain, Dose 1 | 69 | 77
  Grade 3 Pain, Dose 1 | 1 | 2
  Any Redness, Dose 1 | 88 | 86
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 33 | 42
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 420 | 421
  Any Pain, Dose 2 | 47 | 48
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Pain, Dose 2 | 1 | 4
  Any Redness, Dose 2: number analyzed (Participants) | 420 | 421
  Any Redness, Dose 2 | 61 | 66
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 420 | 421
  Any Swelling, Dose 2 | 32 | 27
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Swelling, Dose 2 | 0 | 1
  Any Pain, Across Doses | 89 | 98
  Grade 3 Pain, Across Doses | 2 | 4
  Any Redness, Across Doses | 106 | 106
  Grade 3 Redness, Across Doses | 0 | 0
  Any Swelling, Across Doses | 50 | 51
  Grade 3 Swelling, Across Doses | 0 | 1

36. Secondary Outcome: Number of Subjects Aged 6 Months to <5 Years, Reporting Fever ≥38ºC (100.4°F) and >39.0°C (102.2ºF) Across Doses.
Description: Any fever = all subjects with a documented temperature of ≥ 38°C/100.4°F by any route and all subjects reporting temperature < 38°C but with missing values (MC) for at least one day during the solicited period. Grade 3 fever = temperature above 39.0°C/102.2ºF.
  Data of 2 independent groups were pooled.
Time Frame: During the 2 days (Day 0-Day 1) post-vaccination period
Population: The analysis was performed on the Pediatric-Total Vaccinated cohort which included all subjects aged 6 months to <5 years, with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Groups:
- Influsplit Tetra_IP 6m-<5y Group: Subjects in the Influsplit Tetra_IP group aged between 6 months to <5 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Influsplit Tetra™ vaccine produced by IP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
- Influsplit Tetra_LP 6m-<5y Group: Subjects in the Influsplit Tetra_LP group aged between 6 months to <5 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Influsplit Tetra™ vaccine produced by LP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
Arm/Group | Influsplit Tetra_IP 6m-<5y Group | Influsplit Tetra_LP 6m-<5y Group
Number analyzed (Participants) | 532 | 542
Subjects
  Any Fever | 29 | 31
  Fever (≥38°C) | 28 | 31
  Grade 3 Fever | 4 | 1

37. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were drowsiness, irritability/fussiness, loss of appetite and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 irritability/fussiness was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Grade 3 drowsiness was defined as drowsiness that prevented normal activity. Any fever was defined as subjects with a documented temperature of greater than or equal to (≥) 38°C/100.4°F by any route and all subjects reporting temperature less than (< )38°C but with missing values (MC) for at least one day during the solicited period. Grade 3 fever was defined as temperature greater than (>)39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 462 | 470
Subjects
  Any Drowsiness, Dose 1 | 87 | 77
  Grade 3 Drowsiness, Dose 1 | 3 | 7
  Related Drowsiness, Dose 1 | 54 | 50
  Any Irritability, Dose 1 | 124 | 96
  Grade 3 Irritability, Dose 1 | 10 | 10
  Related Irritability, Dose 1 | 75 | 58
  Any Loss of appetite, Dose 1 | 94 | 76
  Grade 3 Loss of appetite, Dose 1 | 9 | 8
  Related Loss of appetite, Dose 1 | 47 | 40
  Any Fever, Dose 1 | 42 | 44
  Fever (≥38.0°C), Dose 1 | 39 | 42
  Grade 3 Fever, Dose 1 | 8 | 5
  Related Fever, Dose 1 | 16 | 23
  ≥38.0°C Related Fever, Dose 1 | 14 | 22
  Any Drowsiness, Dose 2: number analyzed (Participants) | 420 | 421
  Any Drowsiness, Dose 2 | 63 | 58
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Drowsiness, Dose 2 | 6 | 7
  Related Drowsiness, Dose 2: number analyzed (Participants) | 420 | 421
  Related Drowsiness, Dose 2 | 46 | 35
  Any Irritability, Dose 2: number analyzed (Participants) | 420 | 421
  Any Irritability, Dose 2 | 87 | 87
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Irritability, Dose 2 | 5 | 8
  Related Irritability, Dose 2: number analyzed (Participants) | 420 | 421
  Related Irritability, Dose 2 | 59 | 50
  Any Loss Of Appetite, Dose 2: number analyzed (Participants) | 420 | 421
  Any Loss Of Appetite, Dose 2 | 64 | 69
  Grade 3 Loss Of Appetite, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Loss Of Appetite, Dose 2 | 4 | 10
  Related Loss Of Appetite, Dose 2: number analyzed (Participants) | 420 | 421
  Related Loss Of Appetite, Dose 2 | 39 | 37
  Any Fever, Dose 2: number analyzed (Participants) | 420 | 421
  Any Fever, Dose 2 | 41 | 40
  Fever (≥38.0°C), Dose 2: number analyzed (Participants) | 420 | 421
  Fever (≥38.0°C), Dose 2 | 40 | 40
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Fever, Dose 2 | 10 | 9
  Related Fever, Dose 2: number analyzed (Participants) | 420 | 421
  Related Fever, Dose 2 | 19 | 17
  ≥38.0°C Related Fever, Dose 2: number analyzed (Participants) | 420 | 421
  ≥38.0°C Related Fever, Dose 2 | 19 | 17
  Any Drowsiness, Across Doses | 115 | 103
  Grade 3 Drowsiness, Across Doses | 8 | 13
  Related Drowsiness, Across Doses | 78 | 66
  Any Irritability, Across Doses | 155 | 141
  Grade 3 Irritability, Across Doses | 15 | 17
  Related Irritability, Across Doses | 98 | 87
  Any Loss Of Appetite, Across Doses | 127 | 116
  Grade 3 Loss Of Appetite, Across Doses | 13 | 17
  Related Loss Of Appetite, Across Doses | 69 | 61
  Any Fever, Across Doses | 76 | 70
  Fever (≥38.0°C), Across Doses | 72 | 69
  Grade 3 Fever, Across Doses | 18 | 14
  Related Fever, Across Doses | 32 | 35
  ≥38.0°C Related Fever, Across Doses | 30 | 34

38. Secondary Outcome: Duration of Solicited Local AEs in Subjects Aged 6-35 Months.
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 16
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 88 | 86
Days
  Pain, Dose 1: number analyzed (Participants) | 69 | 77
  Pain, Dose 1 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 7.0]
  Pain, Dose 2: number analyzed (Participants) | 47 | 48
  Pain, Dose 2 | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 6.0]
  Redness, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Redness, Dose 2: number analyzed (Participants) | 61 | 66
  Redness, Dose 2 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Swelling, Dose 1: number analyzed (Participants) | 33 | 42
  Swelling, Dose 1 | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 7.0]
  Swelling, Dose 2: number analyzed (Participants) | 32 | 27
  Swelling, Dose 2 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]

39. Secondary Outcome: Duration of Solicited General AEs in Subjects Aged 6-35 Months.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 16
Measure: Median (Full Range); unit: Days
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 124 | 96
Days
  Drowsiness, Dose 1: number analyzed (Participants) | 87 | 77
  Drowsiness, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 63 | 58
  Drowsiness, Dose 2 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Irritability, Dose 2: number analyzed (Participants) | 87 | 87
  Irritability, Dose 2 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of appetite, Dose 1: number analyzed (Participants) | 94 | 76
  Loss of appetite, Dose 1 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of appetite, Dose 2: number analyzed (Participants) | 64 | 69
  Loss of appetite, Dose 2 | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Fever, Dose 1: number analyzed (Participants) | 42 | 44
  Fever, Dose 1 | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 4.0]
  Fever, Dose 2: number analyzed (Participants) | 41 | 40
  Fever, Dose 2 | 1.0 [1.0 to 5.0] | 2.0 [1.0 to 5.0]

40. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting Solicited Oculorespiratory Syndrome (ORS) Like Symptoms.
Description: as for outcome 12
Time Frame: During a 3 day (Days 0-2) follow-up period after vaccination
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 462 | 470
Subjects
  Any Chest Tightness, Dose 1 | 2 | 1
  Grade 3 Chest Tightness, Dose 1 | 0 | 0
  Related Chest Tightness, Dose 1 | 0 | 0
  Any Cough, Dose 1 | 47 | 50
  Grade 3 Cough, Dose 1 | 3 | 3
  Related Cough, Dose 1 | 16 | 13
  Any Difficulty Breathing, Dose 1 | 15 | 12
  Grade 3 Difficulty Breathing, Dose 1 | 1 | 1
  Related Difficulty Breathing, Dose 1 | 4 | 2
  Any Hoarseness, Dose 1 | 13 | 11
  Grade 3 Hoarseness, Dose 1 | 0 | 0
  Related Hoarseness, Dose 1 | 1 | 4
  Any Red Eyes, Dose 1 | 10 | 11
  Grade 3 Red Eyes, Dose 1 | 0 | 0
  Related Red Eyes, Dose 1 | 6 | 5
  Any Sore throat, Dose 1 | 6 | 7
  Grade 3 Sore throat, Dose 1 | 0 | 0
  Related Sore throat, Dose 1 | 1 | 3
  Any Swallowing Difficulty, Dose 1 | 1 | 5
  Grade 3 Swallowing Difficulty, Dose 1 | 0 | 0
  Related Swallowing Difficulty, Dose 1 | 0 | 2
  Any Swelling of the face, Dose 1 | 4 | 3
  Grade 3 Swelling of the face, Dose 1 | 0 | 0
  Related Swelling of the face, Dose 1 | 1 | 1
  Any Wheezing, Dose 1 | 9 | 12
  Grade 3 Wheezing, Dose 1 | 1 | 1
  Related Wheezing, Dose 1 | 3 | 3
  Any Chest Tightness, Dose 2: number analyzed (Participants) | 420 | 421
  Any Chest Tightness, Dose 2 | 9 | 4
  Grade 3 Chest Tightness, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Chest Tightness, Dose 2 | 0 | 2
  Related Chest Tightness, Dose 2: number analyzed (Participants) | 420 | 421
  Related Chest Tightness, Dose 2 | 0 | 1
  Any Cough, Dose 2: number analyzed (Participants) | 420 | 421
  Any Cough, Dose 2 | 37 | 53
  Grade 3 Cough, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Cough, Dose 2 | 5 | 3
  Related Cough, Dose 2: number analyzed (Participants) | 420 | 421
  Related Cough, Dose 2 | 8 | 8
  Any Difficulty Breathing, Dose 2: number analyzed (Participants) | 420 | 421
  Any Difficulty Breathing, Dose 2 | 19 | 18
  Grade 3 Difficulty Breathing, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Difficulty Breathing, Dose 2 | 1 | 2
  Related Difficulty Breathing, Dose 2: number analyzed (Participants) | 420 | 421
  Related Difficulty Breathing, Dose 2 | 5 | 3
  Any Hoarseness, Dose 2: number analyzed (Participants) | 420 | 421
  Any Hoarseness, Dose 2 | 13 | 9
  Grade 3 Hoarseness, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Hoarseness, Dose 2 | 0 | 1
  Related Hoarseness, Dose 2: number analyzed (Participants) | 420 | 421
  Related Hoarseness, Dose 2 | 1 | 1
  Any Red Eyes, Dose 2: number analyzed (Participants) | 420 | 421
  Any Red Eyes, Dose 2 | 10 | 11
  Grade 3 Red Eyes, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Red Eyes, Dose 2 | 0 | 0
  Related Red Eyes, Dose 2: number analyzed (Participants) | 420 | 421
  Related Red Eyes, Dose 2 | 6 | 1
  Any Sore Throat, Dose 2: number analyzed (Participants) | 420 | 421
  Any Sore Throat, Dose 2 | 7 | 11
  Grade 3 Sore Throat, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Sore Throat, Dose 2 | 1 | 1
  Related Sore Throat, Dose 2: number analyzed (Participants) | 420 | 421
  Related Sore Throat, Dose 2 | 0 | 2
  Any Swallowing Difficulty, Dose 2: number analyzed (Participants) | 420 | 421
  Any Swallowing Difficulty, Dose 2 | 8 | 7
  Grade 3 Swallowing Difficulty, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Swallowing Difficulty, Dose 2 | 2 | 1
  Related Swallowing Difficulty, Dose 2: number analyzed (Participants) | 420 | 421
  Related Swallowing Difficulty, Dose 2 | 0 | 1
  Any Swelling of the face, Dose 2: number analyzed (Participants) | 420 | 421
  Any Swelling of the face, Dose 2 | 5 | 4
  Grade 3 Swelling of the face, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Swelling of the face, Dose 2 | 0 | 0
  Related Swelling of the face, Dose 2: number analyzed (Participants) | 420 | 421
  Related Swelling of the face, Dose 2 | 1 | 1
  Any Wheezing, Dose 2: number analyzed (Participants) | 420 | 421
  Any Wheezing, Dose 2 | 11 | 16
  Grade 3 Wheezing, Dose 2: number analyzed (Participants) | 420 | 421
  Grade 3 Wheezing, Dose 2 | 3 | 1
  Related Wheezing, Dose 2: number analyzed (Participants) | 420 | 421
  Related Wheezing, Dose 2 | 4 | 3
  Any Chest Tightness, Across Doses | 10 | 5
  Grade 3 Chest Tightness, Across Doses | 0 | 2
  Related Chest Tightness, Across Doses | 0 | 1
  Any Cough, Across Doses | 73 | 85
  Grade 3 Cough, Across Doses | 8 | 6
  Related Cough, Across Doses | 22 | 18
  Any Difficulty Breathing, Across Doses | 31 | 25
  Grade 3 Difficulty Breathing, Across Doses | 2 | 3
  Related Difficulty Breathing, Across Doses | 8 | 4
  Any Hoarseness, Across Doses | 23 | 17
  Grade 3 Hoarseness, Across Doses | 0 | 1
  Related Hoarseness, Across Doses | 2 | 5
  Any Red Eyes, Across Doses | 18 | 19
  Grade 3 Red Eyes, Across Doses | 0 | 0
  Related Red Eyes, Across Doses | 10 | 5
  Any Sore Throat, Across Doses | 12 | 17
  Grade 3 Sore Throat, Across Doses | 1 | 1
  Related Sore Throat, Across Doses | 1 | 5
  Any Swallowing Difficulty, Across Doses | 8 | 12
  Grade 3 Swallowing Difficulty, Across Doses | 2 | 1
  Related Swallowing Difficulty, Across Doses | 0 | 3
  Any Swelling of the face, Across Doses | 9 | 7
  Grade 3 Swelling of the face,Across Doses | 0 | 0
  Related Swelling of the face,Across Doses | 2 | 2
  Any Wheezing, Across Doses | 19 | 26
  Grade 3 Wheezing, Across Doses | 4 | 2
  Related Wheezing, Across Doses | 7 | 5

41. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting the Occurrence of All Medically Attended Events (MAEs)
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 466 | 474
Subjects
  Any MAE(s) | 235 | 252
  Grade 3 MAE(s) | 35 | 29
  Related MAE(s) | 2 | 0

42. Secondary Outcome: Number of Subjects Aged 6-35 Months Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 unsolicited AE was defined as an event that prevented normal activity. Related unsolicited AE was defined as an event assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 28-day (Days 0-27) follow-up period after vaccination
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 466 | 474
Subjects
  Any Unsolicited AEs | 243 | 262
  Grade 3 Unsolicited AEs | 33 | 31
  Related Unsolicited AEs | 6 | 3

43. Secondary Outcome: Number of Subjects Aged 6-35 Months, Reporting Any and Related Serious Adverse Events (SAEs)
Description: as for outcome 17
Time Frame: During the entire study period [approximately 28 days (primed subjects) and 56 days (unprimed subjects)]
Population: as for outcome 16
Measure: Number; unit: Subjects
Arm/Group | Influsplit Tetra_IP 6-35m Group | Influsplit Tetra_LP 6-35m Group
Number analyzed (Participants) | 466 | 474
Subjects
  Any SAEs | 7 | 11
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 56; Solicited local and genera l symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: During the 28-day (Days 0-27) post-vaccination period.
Groups:
- Influsplit Tetra_IP 3-17 y: Subjects in the Influsplit Tetra_IP group aged between 3 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by IP at Day 0. Influsplit Tetra™ vaccine produced by IP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
- Influsplit Tetra_LP 3-17 y: Subjects in the Influsplit Tetra_LP group aged between 3 years to <9 years received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Subjects aged 9-17 years received only 1 dose of Influsplit Tetra™ vaccine produced by LP at Day 0. Influsplit Tetra™ vaccine produced by LP was administered intramuscularly in the deltoid region of left or non-dominant arm (Day 0) and in the deltoid region of right or dominant arm (Day 28).
- Influsplit Tetra_IP 6-35 m: Subjects in the Influsplit Tetra_IP group aged between 6 months to 35 months received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by investigational process (IP). Influsplit Tetra™ vaccine produced by IP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
- Influsplit Tetra_LP 6-35 m: Subjects in the Influsplit Tetra_LP group aged between 6 months to 35 months received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Influsplit Tetra™ vaccine produced by licensed process (LP). Influsplit Tetra™ vaccine produced by LP was administered intramuscularly the anterolateral region of left thigh for subjects below 12 months of age and in the deltoid region of left or non-dominant arm in subjects ≥ 12 months of age (Day 0) and in the anterolateral region of right thigh for subjects below 12 months of age and in the deltoid region of right or dominant arm in subjects ≥ 12 months of age (Day 28).
Arm/Group | Influsplit Tetra_IP Adult Group | Influsplit Tetra_LP Adult Group | Influsplit Tetra_IP 3-17 y | Influsplit Tetra_LP 3-17 y | Influsplit Tetra_IP 6-35 m | Influsplit Tetra_LP 6-35 m
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/410 | 0/411 | 0/466 | 0/474
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/60 | 1/410 | 0/411 | 7/466 | 11/474
Other Adverse Events (participants affected / at risk) | 51/60 | 42/60 | 327/410 | 324/411 | 315/466 | 319/474
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influsplit Tetra_IP Adult Group (N=60) | Influsplit Tetra_LP Adult Group (N=60) | Influsplit Tetra_IP 3-17 y (N=410) | Influsplit Tetra_LP 3-17 y (N=411) | Influsplit Tetra_IP 6-35 m (N=466) | Influsplit Tetra_LP 6-35 m (N=474)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pseudocroup (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influsplit Tetra_IP Adult Group (N=60) | Influsplit Tetra_LP Adult Group (N=60) | Influsplit Tetra_IP 3-17 y (N=410) | Influsplit Tetra_LP 3-17 y (N=411) | Influsplit Tetra_IP 6-35 m (N=466) | Influsplit Tetra_LP 6-35 m (N=474)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 35 (36) | 42 (43) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 39 (49) | 56 (64)
Chills (General disorders) | 9 (9) | 7 (7) | 21 (22) | 31 (31) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 43 (46) | 44 (51) | 86 (99) | 100 (124)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 13 (13) | 16 (20) | 127 (158) | 116 (145)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (6) | 13 (13) | 31 (34) | 25 (30)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 131 (145) | 128 (140) | 106 (149) | 107 (153)
Fatigue (General disorders) | 32 (32) | 20 (20) | 97 (102) | 101 (103) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 31 (33) | 37 (44)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (6) | 6 (6) | 38 (38) | 32 (33) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 31 (32) | 16 (17) | 85 (89) | 84 (88) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 10 (11) | 16 (20) | 155 (211) | 141 (183)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (21) | 13 (13) | 72 (74) | 90 (96) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 4 (4) | 6 (6) | 26 (27) | 29 (30)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 16 (17) | 23 (23) | 13 (14) | 18 (20)
Pain (General disorders) | 41 (41) | 32 (32) | 252 (279) | 264 (294) | 89 (117) | 98 (125)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 21 (22) | 24 (25) | 95 (112) | 92 (111)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 16 (19) | 11 (13) | 115 (150) | 103 (135)
Swelling (General disorders) | 2 (2) | 4 (4) | 109 (118) | 110 (117) | 50 (65) | 51 (69)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 13 (14) | 17 (18) | 62 (80) | 73 (82)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 19 (20) | 26 (28)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.